CLINICAL TRIAL: NCT00878111
Title: NGR013: Phase I and Pharmacodynamic Study of NGR-hTNF Administered at High Doses in Patients With Advanced or Metastatic Solid Tumour
Brief Title: Study of NGR-hTNF Administered at High Doses in Patient With Advanced or Metastatic Solid Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR013; 2008-000816-33 (EudraCT Number)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumors
Keywords: NGR-hTNF; Solid tumours; High doses
MeSH Terms: interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: escalating dose levels of NGR-hTNF (Experimental): NGR-hTNF administered at high doses
  Interventions: Drug: NGR-hTNF

INTERVENTIONS:
Drug: NGR-hTNF — First cohort: iv q3W 60 mcg/sqm over 120 min*
  Second cohort: iv q3W 80 mcg/sqm over 120 min*
  Third cohort: iv q3W 100 mcg/sqm over 120 min*
  Fourth cohort: iv q3W 125 mcg/sqm over 120 min*
  Fifth cohort: iv q3W 150 mcg/sqm over 120 min*
  Sixth cohort: iv q3W 175 mcg/sqm over 120 min*
  Seventh cohort: iv q3W 200 mcg/sqm over 120 min*
  Eighth cohort: iv q3W 225 mcg/sqm over 120 min*
  Ninth cohort: iv q3w 250 mcg/sqm over 120 min*
  Tenth cohort: iv q3w 275 mcg/sqm over 120 min*
  Eleventh cohort: iv q3w 300 mcg/sqm over 120 min*
  Twelfth cohort: iv q3w 325 mcg/sqm over 120 min*
  * If the first infusion is well-tolerated, the second infusion may be delivered over 90 minutes. If the 90-minute infusion is well tolerated, all subsequent infusions may be delivered over a 60-minute period.

SUMMARY:
The main objective of the trial is to document the safety and antivascular effect of escalating doses of NGR-hTNF, from 60 mcg/sqm to 325 mcg/sqm, in patients affected by advanced or metastatic solid tumors not amenable of standard therapies.

Safety will be established by clinical and laboratory assessment according to NCI-CTCAE criteria (version 4.02).

DETAILED DESCRIPTION:
Pre-clinical studies provide the support that NGR-TNF is endowed with a higher therapeutic index in animal models and studies of the mechanism of action showed that NGR-TNF can induce tumour necrosis when used at relatively high doses.

Recently, a phase I dose-escalation study of NGR-hTNF has explored the dose range between 0.2 and 60 µg/m2, showing DLT at 60 mcg/m2 experienced as transient acute infusion reaction few minutes after the first administration start. Considering the relationship with the infusion of these events, a further dose escalation will be explored in the present phase I study by using both a longer infusion time (i.e., 120 minutes instead of 60 minutes) and a mild premedication.

The first cohort (n=4) of patients will be treated with NGR-hTNF administered at 60 mcg/m2 IV every three weeks, that is a dose level 33% higher than MTD and recommended dose selected in the previous phase I trial (i.e., 45 mcg/m2). If ≤1 of 4 patients experience DLT during the first cycle, following cohorts will be treated with escalating doses (from 80 to 325 mcg/m2) of NGR-hTNF IV every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with selected metastatic solid tumours recognized to be highly vascularised and not amenable to any clinical improvement by current standard treatments

  * Colorectal cancer (CRC) patients previously resistant to standard systemic regimens (including biologic agents)
  * Gastric cancer (GC) patients treated with no more than two standard systemic regimens for metastatic disease
  * Hepatocellular carcinoma (HCC) patients previously resistant to standard systemic regimens
  * Pancreatic carcinoma (PC) patients treated with no more than one standard systemic regimen for metastatic disease
  * Non small cell lung carcinoma (NSCLC) patients treated with no more than two standard systemic regimens (including biologic agents) for metastatic disease
  * Neuroendocrine (NE) tumours refractory to somatostatin analogue treatment
  * Other rare tumours including malignant pleural mesothelioma (MPM), soft-tissue sarcoma (STS), and renal cell carcinoma (RCC), resistant/refractory to current standard treatments
* Life expectancy more than 3 months
* ECOG Performance status 0-1
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils >1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin <1.5 x ULN
  * AST and/or ALT <2.5 x ULN in absence of liver metastasis
  * AST and/or ALT <5 x ULN in presence of liver metastasis
  * Serum creatinine <1.5 x ULN
  * Creatinine clearance (estimated according to Cockcroft-Gault formula) ≥ 50 ml/min
* Patients may have had prior therapy providing the following conditions are met before treatment start:

  * Chemotherapy, radiation therapy, hormonal therapy, or immunotherapy: wash-out period of 28 days
  * Surgery: wash-out period of 14 days
* Patients must give written informed consent to participate in the study.

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients must not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension
* Prolonged QTc interval (congenital or acquired) > 450 ms
* Patient with significant peripheral vascular disease
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., primary brain tumor, any brain metastasis, seizure not controlled with standard medical therapy), or history of stroke
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of child-bearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Optimal Biologic Dose (OBD) | Before treatment, every 3-6 weeks and at the end of treatment
  Evaluating both the safety in terms of maximum tolerated dose (MTD) and the antivascular effect in terms of changes documented with dynamic imaging (DCE-MRI)

SECONDARY OUTCOMES:
Pharmacokinetic | Several time points after 1st, 2nd and 3rd administration
  Evaluation of plasma levels of sTNF-RI and sTNF-RII and anti-NGR-hTNF antibodies
Preliminary antitumor activity | Every 6 weeks
  In terms of objective response rate according to RECIST criteria, progression-free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy